CLINICAL TRIAL: NCT01341535
Title: A Two-arm Phase II Randomized Study, Comparing Adaptive Biological Imaging - Voxel Intensity - Based Radiotherapy (Adaptive Dose Escalation) Versus Standard Radiotherapy for Head and Neck Cancer.
Brief Title: Comparison of Adaptive Dose Painting by Numbers With Standard Radiotherapy for Head and Neck Cancer.
Acronym: C-ART-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/567
Record Dates: First submitted 2011-04-11; First posted 2011-04-25 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Primary Non-operated Squamous Cell Carcinoma of Oral Cavity; Primary Non-operated Squamous Cell Carcinoma of Oropharynx; Primary Non-operated Squamous Cell Carcinoma of Hypopharynx; Primary Non-operated Squamous Cell Carcinoma of Larynx

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- adaptive DPBN (Experimental): This patient group will be treated by adaptive dose-painting-by-numbers, while patients in the control arm will receive standard treatment.
  Patients will have a 50 % chance of being allocated to the experimental arm and a 50 % chance of being allocated to the control arm.
  Interventions: Radiation: Adaptive dose-painting-by-numbers
- standard IMRT (Active Comparator): This patient group will be treated by standard intensity-modulated radiotherapy (IMRT), while patients in the experimental arm will receive adaptive dose-painting-by-numbers.
  Patients will have a 50 % chance of being allocated to the experimental arm and a 50 % chance of being allocated to the control arm.
  Interventions: Radiation: standard intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Radiation: Adaptive dose-painting-by-numbers — Adaptive dose escalation by dose-painting-by-numbers.
  Arms: adaptive DPBN
Radiation: standard intensity-modulated radiotherapy (IMRT) — Standard radiotherapy for head and neck cancer.
  Arms: standard IMRT

SUMMARY:
The investigators hypothesize that treatment adaptation to biological and anatomical changes, occurring during treatment, can increase the chance of cure at minimized or equal radiation-induced toxicity in head and neck cancer patients. This trial compares standard intensity-modulated radiotherapy (IMRT), using only pre-treatment planning 18F-2-fluoro-2-deoxy-D-glucose positron emission tomography to adaptive 18F-2-fluoro-2-deoxy-D-glucose positron emission tomography voxel intensity based IMRT or volumetric-modulated arc therapy (VMAT) using repetitive per-treatment planning 18F-2-fluoro-2-deoxy-D-glucose positron emission tomography for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of oral cavity, oropharynx, hypopharynx or larynx
* Primary unresectable tumor and/or patients that refused surgery
* Stages T1-4; T3-4 N0 or T(any) N1-3 for glottic cancer
* Multidisciplinary decision of curative radiotherapy or radiochemotherapy
* Karnofsky performance status >= 70 %
* Age >= 18 years old
* Informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* High risk Human Papilloma Virus (HPV)
* Treatment combined with brachytherapy
* Prior irradiation to the head and neck region
* History of prior malignancies, except for cured non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years.
* Distant metastases
* Pregnant or lactating women
* Creatinine clearance (Cockcroft-Gault) =< 60 mL/min
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
To obtain 25 % increase in local control at 1 year with adaptive dose escalation comparing to standard treatment. | at 1 year
  18F-FDG-PET/CT scans will be performed.

SECONDARY OUTCOMES:
Regional (elective neck) and distant control. | after 1 year
  18F-FDG-PET/CT scans will be performed.
Topography of local and/or regional relapse. | during the first year post-treatment
  18F-FDG-PET/CT scans will be performed during the first year post-treatment time point of local and/or regional relapse
Tumor response | 3 months post-treatment
  18F-FDG-PET/CT scans will be performed
Acute toxicity | up to 12 months of follow-up
Overall disease-specific, disease-free survival. | at 1 year
Late toxicity | up to 12 months of follow-up
Time point of local and/or regional relapse. | during the first year post-treatment
  18F-FDG-PET/CT scans will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, Ph.D., M.D., Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Department of Radiotherapy, University Hospital Ghent, Ghent
  - Clinique & Materinité Sainte Elisabeth, Namur

REFERENCES:
- See also: Related Info — http://www.uzgent.be